CLINICAL TRIAL: NCT07158931
Title: Investigation of Effectiveness of 'Nordic Walking' Training On Geriatric Individuals: a Randomized Comparative Study
Brief Title: 'Nordic Walking' on Geriatric Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Rumeli University (Other)
Responsible Party: Principal Investigator, Nursel Oziri, PhD, Istanbul Rumeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulRumeliU
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Geriatrics; Geriatric Rehabilitation
MeSH Terms: interventions — Nordic Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Nordic Walking
  Interventions: Other: nordic walking
- Control (Active Comparator): General walking
  Interventions: Other: General walking

INTERVENTIONS:
Other: nordic walking — Before the NW program, participants completed a one-week familiarization phase to practice pole use. Training was held three times: 15 minutes on days 1 and 2, and 20 minutes on day 3, at 40-60% heart rate reserve (measured with a pulse oximeter). Warm-up included a 1-minute slow walk, toe raises, seated dorsiflexion, mini squats, scapular adduction, and shoulder/wrist stretches. Each session ended with a cool-down of a 2-minute slow walk and 20-second stretches for major muscle groups (quadriceps, hamstrings, lumbar extensors, gastrocnemius, shoulders, wrists).The walking poles used in this study were the Evolite Ultralite Titanium Antishock Trekking Pole, which has a titanium alloy body and a three-piece telescopic structure, adjustable to the desired length between 68 and 135 cm.
  Arms: Experimental
Other: General walking — The program was performed on concrete or compacted soil surfaces, under the same physiotherapist's supervision. Walking speed was adjusted to remain below 60% of maximal heart rate and to allow participants to converse comfortably during exercise.
  Arms: Control

SUMMARY:
This study aimed to investigate the effects of Nordic Walking training on muscle strength and endurance, balance, fear of falling, aerobic capacity, fatigue, quality of life and activity level in geriatric individuals.

32 sedentary individuals between the ages of 65-80 participated in the study. Nordic Walking (NW) and Traditional Walking (GY) groups were created by systematic randomization method. In line with the intended research parameters, participants were given 30 sec sit-to-stand (30secCST), 30 sec biceps curl (30 sec ACT), timed up and go (TUG) 6 min walk (6MWT), Tinetti Fall Effectiveness (Tinetti FES), Tampa Kinesiophobia Scale (TSK), World Health Organization Quality of Life Elderly Module (WHOQOL-Old) were administered. Evaluations were repeated before and after the study. The study was conducted under the supervision of a physiotherapist, 3 days a week for 12 weeks in both groups.

ELIGIBILITY:
Inclusion Criteria:

* being between 65 and 80 years of age,
* having a score of 24 or above on the Standardized Mini-Mental State Examination (SMMSE),
* and voluntarily agreeing to participate in the study.

Exclusion Criteria:

* a history of cerebrovascular accident,
* acute retinal hemorrhage or previous ophthalmic surgery,
* active infection, malignancy,
* multiple organ failure, terminal illness, or a history of lower or upper extremity fracture within the last three months.
* had any musculoskeletal condition that would prevent them from engaging in exercise,
* a diagnosis of Alzheimer's disease, Parkinson's disease, or dementia,
* a diagnosis of benign paroxysmal positional vertigo (BPPV),
* had engaged in regular exercise training (≥150 minutes per week) within the past six months.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Sit-to-stand test (STS): | at the beginning and at the end of the 12th week
  This is a widely used clinical assessment tool in geriatrics for evaluating lower limb function, muscle strength, balance, and overall physical performance in older adults. Participants were instructed to sit on a chair approximately 48 cm in height, keeping their back straight, feet flat on the floor, and arms crossed over the chest. They were then asked to stand up and sit down repeatedly for 30 seconds. The total number of complete stands performed within the 30-second period was recorded
Biceps curl test (BCT): | at the beginning and at the end of the 12th week
  This is a widely used assessment in geriatrics to evaluate upper body strength and endurance, particularly of the arm muscles (7). The arm curl test was performed with participants seated on a chair without armrests. Holding a dumbbell in the hand with the palm facing the body, participants executed elbow flexion with supination through a full range of motion, ensuring the elbow was fully bent and then fully extended for each repetition. Women used 2 kg dumbbells and men used 3 kg dumbbells. The total number of controlled repetitions completed in 30 seconds was recorded.
6-Minute Walk Test (MWT): | at the beginning and at the end of the 12th week
  It is a widely used, simple, and validated clinical assessment to measure aerobic capacity and functional exercise tolerance in older adults (8). The participant was instructed to walk along a 30-meter flat surface for six minutes. At the end of the six-minute period, the total distance walked was recorded in meters.
Timed Up and Go Test (TUG): | at the beginning and at the end of the 12th week
  This is a clinical and research tool to assess mobility, balance, walking ability, and fall risk in older adults (9). While seated on a chair approximately 48 cm in height, the participant was instructed, upon hearing the "start" command, to stand up, walk 3 meters forward at a normal walking speed, return, and sit down again. The test was performed twice, and the average time was recorded.

SECONDARY OUTCOMES:
Tinetti Falls Efficacy Scale (TFES): | at the beginning and at the end of the 12th week
  It is a validated tool used to assess an individual's confidence in performing daily activities without falling. Participants rated their perceived safety during various daily activities on a scale from 1 (very confident) to 10 (not confident at all). Scores were converted to a total between 0 (low fall-related self-efficacy) and 100 (high fall-related self-efficacy), with higher scores indicating greater fear of falling (10).
Tampa Kinesiophobia Scale (TKS): | at the beginning and at the end of the 12th week
  It is a 17-item self-report questionnaire rated on a 4-point Likert scale, designed to assess fear of movement or re-injury. Higher scores indicate greater levels of kinesiophobia.
World Health Organization Quality of Life Instrument-Older Adults Module (WHOQL- OLD): | at the beginning and at the end of the 12th week
  It is a 24-item questionnaire assessed on a five-point Likert scale, covering six domains: sensory abilities, autonomy, past-present-future activities, social participation, death and dying, and intimacy. Each domain is scored from 4 to 20, and higher total scores indicate better quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Öziri, Ataşehir, Istanbul, Turkey (Türkiye)